CLINICAL TRIAL: NCT01389154
Title: A Pilot Prospective Study Evaluating the SPiN Drive(TM)Electromagnetic Tip Tracked Devices Used in Diagnostic Bronchoscopy
Brief Title: Pilot Study to Measure Lung Biopsy Diagnostic Yield Using Always On Electromagnetic Tip Tracked Devices
Acronym: ALOSPNDY
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Product Enhancements completed
Sponsor: Veran Medical Technologies (Industry)
Collaborators: Institute for Quality Resource Management (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: VMT-SPiN_01
Record Dates: First submitted 2011-07-01; First posted 2011-07-07 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Coin Lesion
Keywords: diagnostic yield; Electromagnetic Tip Tracked; peripheral lung lesion
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients recommended for a lung biopsy. (Experimental): Patients with a positive diagnosis of a peripheral, less than 3.0 centimeter lung lesion, recommended for bronchoscopic biopsy are eligible to be consented into the study.
  Interventions: Procedure: Lung biopsy using Always On EM Tip Tracked Device

INTERVENTIONS:
Procedure: Lung biopsy using Always On EM Tip Tracked Device — Patients screened by CT to have a subsegmental, less than 3.0 centimeter lung lesion will be assigned to outpatient bronchoscopy. The patient will have a chest CT with the Always on Patient vPad. Access to the lesion will be achieved using Electromagnetic Tip Tracked devices. Once accessed the operator will use the Electromagnetic Tip Tracked devices or standard devices to obtain a biopsy sample to then be to pathology for diagnosis and reporting. Once completed the patient will be moved to recovery and discharged. If the biopsy is negative the patient will be advised by the pulmonologist about other interventions, watchful waiting, or no further treatment. If the biopsy is positive, the patient will be referred to their physician for further treatment.
  Other Names: Always On Electromagnetic Tip Tracked Diagnostic Yield

SUMMARY:
The objective of the prospective, multi-center study is to evaluate the ease of use and effectiveness of the SPiN Drive Electromagnetic (EM) Tip Tracked Steerable Devices as a method of sampling subsegmental, less than 3.0 cm, lung lesions through the airway, and beyond the bronchus. Measures of diagnostic yield will be compared to the diagnostic yield of similar published historical controls using conventional bronchoscopy.

DETAILED DESCRIPTION:
Always On EM Tip Tracked Steerable catheters and biopsy devices used with the Veran Medical Technologies system are Food and Durg Administration 510K approved for use in diagnostic pulmonary procedures to locate and sample subsegmental peripheral, less than 3.0 centimeter lung lesions or solitary pulmonary nodules(SPN).

Up to 20 subjects with radiographically confirmed peripheral lung lesions will be asked to participate in the study and proceed with informed consent. An interim analysis of the data will be conducted to determine the need to include an additional 10 patients to achieve statistically significant results at the ninety five percent confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides informed consent
* Subject is older than 50 years of age with 50% of patients at least 65 years of age
* Patient has a minimum of 20 pack years
* Subject scheduled to undergo conventional bronchoscopy as part of their standard medical care
* Subject has radiographically confirmed sub-segmental peripheral < 3.0 cm lung lesions
* A negative pregnancy test in women of child-bearing potential
* Subject is willing and able to return for all required follow-up
* Subject is mentally capable of following study directions

Exclusion Criteria:

* Subject has pacemaker, implantable cardioverter, and/or defibrillator
* Subject has any disease or condition that interferes with safe completion of initial or follow-up assessments
* Pregnant or nursing female subjects, or female subjects of child bearing potential who refuse to take a pregnancy prior to their enrollment in this study
* Concurrent participation in another study involving investigational drugs or investigational medical devices
* Inability to read and understand the necessary study documents

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of a subsegmental pulmonary lesion of less than 3.0 cm. | Within 1 week
  Biopsy samples will be sent to the lab for analysis of the presence, absence, or identification of an occult particulate taken from the patient's lung. Patients with a negative biopsy result will be followed if recommended for another intervention and if recommended to watchful waiting. Follow up outcomes will be included in the outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Momen Wahidi, MD, MBA, Principal Investigator — Duke University

REFERENCES:
- [Background] Schreiber G, McCrory DC. Performance characteristics of different modalities for diagnosis of suspected lung cancer: summary of published evidence. Chest. 2003 Jan;123(1 Suppl):115S-128S. doi: 10.1378/chest.123.1_suppl.115s. PMID 12527571
- [Background] Reichenberger F, Weber J, Tamm M, Bolliger CT, Dalquen P, Perruchoud AP, Soler M. The value of transbronchial needle aspiration in the diagnosis of peripheral pulmonary lesions. Chest. 1999 Sep;116(3):704-8. doi: 10.1378/chest.116.3.704. PMID 10492275
- [Background] Tan BB, Flaherty KR, Kazerooni EA, Iannettoni MD; American College of Chest Physicians. The solitary pulmonary nodule. Chest. 2003 Jan;123(1 Suppl):89S-96S. doi: 10.1378/chest.123.1_suppl.89s. PMID 12527568
- [Background] Alberg AJ, Samet JM. Epidemiology of lung cancer. Chest. 2003 Jan;123(1 Suppl):21S-49S. doi: 10.1378/chest.123.1_suppl.21s. PMID 12527563
- [Background] Edell E, Krier-Morrow D. Navigational bronchoscopy: overview of technology and practical considerations--new Current Procedural Terminology codes effective 2010. Chest. 2010 Feb;137(2):450-4. doi: 10.1378/chest.09-2003. Epub 2009 Dec 4. PMID 19965952
- [Background] Herth FJ, Eberhardt R, Becker HD, Ernst A. Endobronchial ultrasound-guided transbronchial lung biopsy in fluoroscopically invisible solitary pulmonary nodules: a prospective trial. Chest. 2006 Jan;129(1):147-50. doi: 10.1378/chest.129.1.147. PMID 16424425
- [Background] Shirakawa T, Imamura F, Hamamoto J, Honda I, Fukushima K, Sugimoto M, Shirkakusa T. Usefulness of endobronchial ultrasonography for transbronchial lung biopsies of peripheral lung lesions. Respiration. 2004 May-Jun;71(3):260-8. doi: 10.1159/000077424. PMID 15133346
- [Background] Landi S, Cenni MC, Maffei L, Berardi N. Environmental enrichment effects on development of retinal ganglion cell dendritic stratification require retinal BDNF. PLoS One. 2007 Apr 4;2(4):e346. doi: 10.1371/journal.pone.0000346. PMID 17406670
- [Background] Makris D, Scherpereel A, Leroy S, Bouchindhomme B, Faivre JB, Remy J, Ramon P, Marquette CH. Electromagnetic navigation diagnostic bronchoscopy for small peripheral lung lesions. Eur Respir J. 2007 Jun;29(6):1187-92. doi: 10.1183/09031936.00165306. Epub 2007 Mar 14. PMID 17360724
- [Background] Eberhardt R, Anantham D, Ernst A, Feller-Kopman D, Herth F. Multimodality bronchoscopic diagnosis of peripheral lung lesions: a randomized controlled trial. Am J Respir Crit Care Med. 2007 Jul 1;176(1):36-41. doi: 10.1164/rccm.200612-1866OC. Epub 2007 Mar 22. PMID 17379850
- [Background] Gildea TR, Mazzone PJ, Karnak D, Meziane M, Mehta AC. Electromagnetic navigation diagnostic bronchoscopy: a prospective study. Am J Respir Crit Care Med. 2006 Nov 1;174(9):982-9. doi: 10.1164/rccm.200603-344OC. Epub 2006 Jul 27. PMID 16873767
- [Background] Lamprecht B, Porsch P, Pirich C, Studnicka M. Electromagnetic navigation bronchoscopy in combination with PET-CT and rapid on-site cytopathologic examination for diagnosis of peripheral lung lesions. Lung. 2009 Jan-Feb;187(1):55-9. doi: 10.1007/s00408-008-9120-8. Epub 2008 Oct 5. PMID 18836886
- [Background] Schwarz Y, Greif J, Becker HD, Ernst A, Mehta A. Real-time electromagnetic navigation bronchoscopy to peripheral lung lesions using overlaid CT images: the first human study. Chest. 2006 Apr;129(4):988-94. doi: 10.1378/chest.129.4.988. PMID 16608948
- [Background] Hautmann H, Schneider A, Pinkau T, Peltz F, Feussner H. Electromagnetic catheter navigation during bronchoscopy: validation of a novel method by conventional fluoroscopy. Chest. 2005 Jul;128(1):382-7. doi: 10.1378/chest.128.1.382. PMID 16002960
- See also: Reduced Lung-Cancer Mortality with Low-Dose CT Screening — http://www.nejm.org/doi/pdf/10.1056/NEJMoa1102873